CLINICAL TRIAL: NCT03468972
Title: Effect of Immunosuppression in IgA Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0303
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Biopsy-proven IgA Nephropathy
Keywords: IgA nephropathy; immunosuppression
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunosuppression (Experimental): corticosteroids or cyclophosphamide added on corticosteroids
  Interventions: Drug: Immunosuppressive treatment
- Intensive supportive care (Active Comparator): intensive supportive care with RAS blockers, blood pressure control, and protein restriction diet
  Interventions: Other: intensive supportive care

INTERVENTIONS:
Drug: Immunosuppressive treatment — At 3 months after randomization, patients in the corticosteroid arm who have persistent proteinuria of ≥ 1.0 g/g creatinine, or fast decline in eGFR ≥ 15% from the baseline value, will additionally receive cyclosphosphamide during the following 3 months. Patients who have substantial decreased amount of proteinuria < 1.0 g/g creatinine at 3 months will continue protocol-based corticosteroids during the same period. At 6 months after randomization, patients who receive add-on cyclophosphamide will switch to azathioprine as a maintenance therapy and those who receive corticosteroids alone will discontinue the treatment and will be followed up during 24 months thereafter. Assessment of outcome will be done at 6 months and at 36 months.
  Arms: Immunosuppression
Other: intensive supportive care — During 3-6 months before the enrollment, all patients will receive maximal supportive care including the use of RAS blockers, blood pressure control with a target of <130/80 mmHg, and protein restriction diet. If proteinuria does not decrease < 1.0 g/g creatinine, patients will be randomly assigned to continue supportive care, or to receive corticosteroids.
  Arms: Intensive supportive care

SUMMARY:
IgA nephropathy (IgAN) is the most common glomerulonephritis worldwide, leading to end stage renal disease (ESRD) in up to 30 to 40% of patients with in a few decades after diagnosis. Several therapeutic options have been used in clinical practice. However, no treatments can completely stop the progression of IgAN. Given the pathogenic mechanism of IgAN, many researchers have tried to treat patients with IgAN using immunosuppression such as corticosteroids. To date, there have been conflicting results on the effects of immunosuppression in IgAN. Earlier studies from Italian groups showed that corticosteroid treatment significantly attenuated kidney function decline and decreased the development of ESRD. Since then, the beneficial effects of corticosteroids have generally been accepted for treatment of IgAN particularly in patients with high degree of proteinuria > 1.0 g/day despite maximal conservative care during 3 to 6 months. However, a recent interventional study by German group, known as the Supportive Versus Immunosuppressive Therapy for the Treatment of Progressive IgA Nephropathy (STOP-IgAN) trial, showed that immunosuppressive treatment in addition to intensive supportive care did not significantly improve renal outcome and resulted in more treatment-related side effects. Moreover, the Therapeutic Evaluation of Steroids in IgA Nephropathy Global (TESTING) study, another randomized controlled study from China, was early terminated because of safety concern related to corticosteroids. Interestingly, the primary composite outcome occurred significantly less in the methylprednisolone group as compared to the placebo group despite more serious adverse events in the former group. With this background in mind, we designed a multicenter prospective randomized controlled open-label trial; a step-wise therapeutic approach with corticosteroids or add-on cyclophosphamide therapy in IgAN patients with persistent proteinuria who have preserved eGFR of ≥ 30 ml/min/1.73 m2. A total of 19 hospitals will participate in this study. During 12 weeks before the enrollment, all patients will receive maximal supportive care including the use of RAS blockers, blood pressure control with a target of <130/80 mmHg, and protein restriction diet. If proteinuria does not decrease < 1.0 g/g creatinine, patients will be randomly assigned to continue supportive care, or to receive corticosteroids. At 3 months after randomization, patients in the corticosteroid arm who have persistent proteinuria of ≥ 1.0 g/g creatinine, or fast decline in eGFR ≥ 15% from the baseline value, will additionally receive cyclosphosphamide during the following 3 months. Patients who have substantial decreased amount of proteinuria < 1.0 g/g creatinine at 3 months will continue protocol-based corticosteroids during the same period. At 6 months after randomization, patients who receive add-on cyclophosphamide will switch to azathioprine as a maintenance therapy and those who receive corticosteroids alone will discontinue the treatment and will be followed up during 24 months thereafter. At least 87 subjects (a total of 174) would be required for each group to detect 13.5% difference in response rates between the two groups based on previous studies if type I error rate is 5% and type II error is 20% given 20% of drop-out rate during the study period. The primary endpoint is the development of a ≥ 30% decline in eGFR from the baseline or the onset of ESRD. This study will unveil conflicting results on the effects of immunosuppressive treatment in IgAN patients at high risk of progression.

DETAILED DESCRIPTION:
The investigators will conduct a multicenter prospective randomized controlled open-label trial; a step-wise therapeutic approach in IgAN patients with persistent proteinuria who have preserved eGFR of ≥ 30 ml/min/1.73 m2. During 3-6 months before the enrollment, all patients will receive maximal supportive care including the use of RAS blockers, blood pressure control with a target of <130/80 mmHg, and protein restriction diet. If proteinuria does not decrease < 1.0 g/g creatinine, patients will be randomly assigned to continue supportive care, or to receive corticosteroids. At 3 months after randomization, patients in the corticosteroid arm who have persistent proteinuria of ≥ 1.0 g/g creatinine, or fast decline in eGFR ≥ 15% from the baseline value, will additionally receive cyclosphosphamide during the following 3 months. Patients who have substantial decreased amount of proteinuria < 1.0 g/g creatinine at 3 months will continue protocol-based corticosteroids during the same period. At 6 months after randomization, patients who receive add-on cyclophosphamide will switch to azathioprine as a maintenance therapy and those who receive corticosteroids alone will discontinue the treatment and will be followed up during 24 months thereafter. At least 87 subjects (a total of 174) would be required for each group to detect 13.5% difference in response rates between the two groups based on previous studies if type I error rate is 5% and type II error is 20% given 20% of drop-out rate during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven IgA nephropathy within 5 years of enrollment
* Persistent proteinuria of UPCR ≥ 1.0 g/g creatinine during 12-week supportive care including RAS blockers
* baseline eGFR ≥ 30 ml/min/1.73 m2 assessed by CKD-EPI equation

Exclusion Criteria:

* Nephrotic syndrome, atypical IgA nephropathy
* Crescents ≥ 25%
* Overt pulmonary tuberculosis
* Malignancy within 5 years of enrollment
* Pregnancy or breast feeding
* Active hepatitis, chronic hepatitis, liver cirrhosis, HIV
* Kidney transplant
* Current use of immunosuppressive treatment or prior use of immunosuppressive drugs within 1 year of enrollment
* Uncontrolled hypertension (> 160/100 mmHg)
* Aged < 19 years
* Secondary IgA nephropathy such as lupus nephritis, chronic liver disease, or Henoch-Schlein purpura
* Involvement of other clinical trials within 3 months of enrollment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
progression of disease | 6 months
  a composite of a ≥ 30% decline in eGFR from the baseline or the onset of ESRD
progression of disease | 36 months
  a composite of a ≥ 30% decline in eGFR from the baseline or the onset of ESRD

SECONDARY OUTCOMES:
Changes in urinary protein excretion and hematuria | 6 months
Changes in urinary protein excretion and hematuria | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Manno C, Torres DD, Rossini M, Pesce F, Schena FP. Randomized controlled clinical trial of corticosteroids plus ACE-inhibitors with long-term follow-up in proteinuric IgA nephropathy. Nephrol Dial Transplant. 2009 Dec;24(12):3694-701. doi: 10.1093/ndt/gfp356. Epub 2009 Jul 23. PMID 19628647
- [Result] Rauen T, Eitner F, Fitzner C, Sommerer C, Zeier M, Otte B, Panzer U, Peters H, Benck U, Mertens PR, Kuhlmann U, Witzke O, Gross O, Vielhauer V, Mann JF, Hilgers RD, Floege J; STOP-IgAN Investigators. Intensive Supportive Care plus Immunosuppression in IgA Nephropathy. N Engl J Med. 2015 Dec 3;373(23):2225-36. doi: 10.1056/NEJMoa1415463. PMID 26630142
- [Result] Lv J, Zhang H, Wong MG, Jardine MJ, Hladunewich M, Jha V, Monaghan H, Zhao M, Barbour S, Reich H, Cattran D, Glassock R, Levin A, Wheeler D, Woodward M, Billot L, Chan TM, Liu ZH, Johnson DW, Cass A, Feehally J, Floege J, Remuzzi G, Wu Y, Agarwal R, Wang HY, Perkovic V; TESTING Study Group. Effect of Oral Methylprednisolone on Clinical Outcomes in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):432-442. doi: 10.1001/jama.2017.9362. PMID 28763548
- [Result] Lv J, Zhang H, Chen Y, Li G, Jiang L, Singh AK, Wang H. Combination therapy of prednisone and ACE inhibitor versus ACE-inhibitor therapy alone in patients with IgA nephropathy: a randomized controlled trial. Am J Kidney Dis. 2009 Jan;53(1):26-32. doi: 10.1053/j.ajkd.2008.07.029. Epub 2008 Oct 19. PMID 18930568
- [Result] Pozzi C, Bolasco PG, Fogazzi GB, Andrulli S, Altieri P, Ponticelli C, Locatelli F. Corticosteroids in IgA nephropathy: a randomised controlled trial. Lancet. 1999 Mar 13;353(9156):883-7. doi: 10.1016/s0140-6736(98)03563-6. PMID 10093981
- [Result] Tesar V, Troyanov S, Bellur S, Verhave JC, Cook HT, Feehally J, Roberts IS, Cattran D, Coppo R; VALIGA study of the ERA-EDTA Immunonephrology Working Group. Corticosteroids in IgA Nephropathy: A Retrospective Analysis from the VALIGA Study. J Am Soc Nephrol. 2015 Sep;26(9):2248-58. doi: 10.1681/ASN.2014070697. Epub 2015 Feb 12. PMID 25677392